CLINICAL TRIAL: NCT06336707
Title: A Phase I Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Efficacy of HS-20089 Combination Treatment in Subjects With Advanced Solid Tumors
Brief Title: HS-20089 Combination Treatment in Subjects With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hansoh BioMedical R&D Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HS-20089-103
Record Dates: First submitted 2024-03-20; First posted 2024-03-29 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Advanced Solid Tumors
Keywords: HS-20089; B7-H4; Antibody-drug Conjugate; Combination Therapy
MeSH Terms: interventions — Bevacizumab; Cisplatin; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- HS-20089 and Adebrelimab (Experimental)
  Interventions: Drug: HS-20089; Drug: Adebrelimab
- HS-20089, Adebrelimab and cisplatin / carboplatin (Experimental)
  Interventions: Drug: HS-20089; Drug: Adebrelimab; Drug: Cisplatin / carboplatin
- HS-20089 and Bevacizumab (Experimental)
  Interventions: Drug: HS-20089; Drug: Bevacizumab
- HS-20089, Bevacizumab and cisplatin / carboplatin (Experimental)
  Interventions: Drug: HS-20089; Drug: Bevacizumab; Drug: Cisplatin / carboplatin

INTERVENTIONS:
Drug: HS-20089 — Intravenous infusion
Drug: Adebrelimab — Intravenous infusion
  Arms: HS-20089 and Adebrelimab; HS-20089, Adebrelimab and cisplatin / carboplatin
Drug: Bevacizumab — Intravenous infusion
  Arms: HS-20089 and Bevacizumab; HS-20089, Bevacizumab and cisplatin / carboplatin
Drug: Cisplatin / carboplatin — Intravenous infusion
  Arms: HS-20089, Adebrelimab and cisplatin / carboplatin; HS-20089, Bevacizumab and cisplatin / carboplatin

SUMMARY:
HS-20089 is an investigational antibody-drug conjugate (ADC) composed of a humanized IgG1 anti-B7-H4 monoclonal antibody conjugated to the topoisomerase I inhibitor payload via a protease-cleavable linker, with an average drug-to-antibody ratio of about 6.

This is a phase Ⅰ, open-label, multi-center study to evaluate the safety, tolerability, pharmacokinetics (PK) and efficacy of HS-20089 in combination with other antitumor agents (Adebrelimab with or without platinum; Bevacizumab with or without platinum) in subjects with advanced solid tumors.

DETAILED DESCRIPTION:
This study contains four combination therapy cohorts, each consisting of a dose exploration part and a dose expansion part.

The dose exploration part will explore the corresponding optimal dose level of HS-20089 in each combination therapy. The dose expansion part will be conducted at 1 or 2 safe and potentially effective dose levels in subjects with selected tumors in each cohort.

The cohorts may be adjusted based on the observed clinical results, translational medicine data and research progress in the field.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females aged 18 years or older (≥18 years).
2. Patients diagnosed with pathologically confirmed advanced solid tumors.
3. Subjects have at least one target lesion as assessed per the RECIST 1.1. Patients with only brain and/or bone lesions as target lesions are ineligible.
4. Agree to provide fresh or archival tumor tissue
5. Eastern Cooperative Oncology Group Performance Status (ECOG PS) score of 0 to 1 and no deterioration within 2 weeks before the first dose.
6. Have a life expectancy of at least 12 weeks.
7. Female subjects of childbearing potential are willing to take appropriate contraceptive measures and should not breastfeed from signing the informed consent until 6 months after the last dose; male subjects must agree to use barrier contraception (i.e. condoms) from signing the informed consent to 6 months after the last dose.
8. Female subjects must have a negative pregnancy test within 7 days prior to the first dose (for subjects with tumor related abnormal elevation of human chorionic gonadotropin [HCG], an ultrasound of uterus and appendages should be performed within 7 days prior to the first dose to rule out pregnancy), or demonstrate no risk for pregnancy.
9. Subject must be voluntarily enrolled in this clinical trial, be able to understand the study procedures and to sign written informed consent.

Exclusion Criteria:

1. Have received or is currently receiving the following treatment: B7-H4-targeted therapies; Have received any of cytotoxic chemotherapy drugs, investigational drugs, anti-tumor traditional Chinese medicines or other anti-tumor drugs within 14 days prior to the first dose of study drug; or need to continue these drugs during the study.
2. Presence of Grade ≥ 2 toxicities as per Common Terminology Criteria for Adverse Events due to prior anti-tumor therapy.
3. Presence of pleural/abdominal effusion requiring clinical intervention.
4. Known history of other primary malignancy.
5. Evidence of brain metastasis and/or cancerous meningitis
6. Inadequate bone marrow reserve or hepatic/renal functions.
7. Cardiological examination abnormality.
8. Severe, uncontrolled or active cardiovascular disorders.
9. Serious or poorly controlled diabetes.
10. Serious or poorly controlled hypertension.
11. Clinically significant bleeding symptoms or significant bleeding tendency within 1 month prior to the first dose of study treatment.
12. Serious infections within 4 weeks prior to the first dose.
13. Have received systemic glucocorticoid therapy for more than 7 days within 28 days prior to the first dose study treatment, or require chronic (≥ 7 days) use of systemic glucocorticoids during the study, or have other acquired, congenital immunodeficiency disorders, or a history of organ transplantation.
14. Presence of active infectious diseases such as hepatitis B, hepatitis C, tuberculosis, syphilis, or human immunodeficiency virus infection, etc.
15. Current hepatic encephalopathy, hepatorenal syndrome, or Child-Pugh Class B or more severe cirrhosis.
16. Any moderate or severe lung diseases that may interfere with the detection and treatment of drug-related pulmonary toxicity or may seriously affect respiratory function.
17. History of severe neurological or psychiatric disorder.
18. Pregnant or breast-feeding women or women who intend to become pregnant during the study.
19. Attenuated live vaccination within 4 weeks prior to the first dose.
20. Subjects with autoimmune disease that is active or is likely to recur.
21. Subjects with gastrointestinal fistula, visceral fistula, gastrointestinal perforation, or abdominal abscess, or with symptoms/signs of intestinal obstruction within 6 months prior to the first dose of study drug.
22. Subjects unlikely to comply with study procedures, restrictions and requirement as determined by the investigator.
23. Subjects with any condition that jeopardizes the safety of the patient or interferes with the assessment of the study, as judged by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1048 (Estimated)
Dates: Start 2024-04-11 (Actual); Primary Completion 2026-04-08 (Estimated); Study Completion 2028-04-08 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) or maximum applicable dose (MAD) of HS-20089 in combination therapy | Up to day 21 from the first dose
  To determine the MTD or MAD of HS-20089 in each combination therapy.

SECONDARY OUTCOMES:
Incidence and severity of adverse events (AEs) | From the first dose to 90 days after the end of treatment
  AEs will be graded according to the NCI Common Terminology Criteria for Adverse Events (CTCAE), Version 5.0. Incidence and severity of AEs are assessed according to vital signs, laboratory variables, physical examination, electrocardiogram, etc.
Observed maximum plasma concentration (Cmax) of HS-20089 | From pre-dose to 14 days after the first dose of HS-20089 on Cycle 1 (each cycle is 21 days).
  Cmax will be obtained following administration of the first dose of HS-20089 during the first cycle.
Time to reach maximum plasma concentration (Tmax) of HS-20089 following the first dose | From pre-dose to 14 days after the first dose on Cycle 1 (each cycle is 21 days).
  Tmax will be obtained following administration of the first dose of HS-20089 during the first cycle.
Area under plasma concentration versus time curve from zero to last sampling time (AUC0-t) following the first dose of HS-20089 | From pre-dose to 14 days after the first dose on Cycle 1 (each cycle is 21 days).
  Area under the plasma concentration versus time curve from time zero to the last sampling time when the concentration is no less than the lower limit of quantification (LLQ). AUC0-t will be calculated according to the mixed log-linear trapezoidal rule.
Area under the plasma concentration versus time curve from time zero to infinity (AUC0-∞) after single dose of HS-20089 | From pre-dose to 14 days after the first dose on Cycle 1 (each cycle is 21 days).
  AUC0-∞ will be calculated by combining AUC0-t and AUCextra. AUCextra represents an extrapolated value obtained by Clast/ λz, where Clast is the calculated plasma concentration at the last sampling time point at which the measured plasma concentration is at or above the LLQ and λz is the apparent terminal rate constant determined by log-linear regression analysis of the measured plasma concentrations of the terminal log-linear phase.
Objective response rate (ORR) assessed by investigators according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 | From the first dose up to disease progression or withdrawal from study, whichever came first (assessed up to 24 months).
  ORR is defined as the percentage of participants who achieved a best overall response (BOR) of confirmed complete response (CR) or partial response (PR), assessed by investigators based on RECIST 1.1.
Duration of response (DoR) assessed by investigators according to RECIST 1.1 | From the first dose to disease progression or withdrawal from study, whichever came first (assessed up to 24 months).
  DoR is defined as the period from the first occurrence of CR or PR to progressive disease (PD) or death of any cause. If no PD or death after CR/PR, the cut-off date of progression-free survival (PFS) will be used.
Disease control rate (DCR) assessed by investigators according to RECIST 1.1 | From the first dose to disease progression or withdrawal from study, whichever came first (assessed up to 24 months).
  DCR is defined as the percentage of participants with BOR of confirmed CR, PR and stable disease (SD).
Progression-free survival (PFS) assessed by investigators according to RECIST 1.1 | From the first dose or randomization to disease progression or withdrawal from study, whichever came first (assessed up to 24 months).
  PFS is defined as the time from first dose or randomization (if any) to PD or death of any cause.
Overall survival (OS) | From the first dose or randomization to death or withdrawal from study, whichever came first, assessed up to 24 months.
  OS is defined as the time from the first dose or randomization (if any) to death of any cause.
Percentage of participants with antibodies to HS-20089 in serum | From the first dose to 90 days after the end of treatment.
  Serum samples will be collected for the determination of anti-drug antibody (ADA) at designated time points.

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital affiliated to Tongji Medical College of Huazhong University of Science & Technology, Shanghai, Shanghai Municipality, China